CLINICAL TRIAL: NCT05875610
Title: Clinical Study on Chemotherapy Induced Peripheral Neuropathy: Preventive Approach Using Venlafaxine
Brief Title: Preventive Approach Using Venlafaxine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mit Ghamr Oncology Center (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahrous Ali, Head of clinical pharmacy department, Mit Ghamr Oncology Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy
Keywords: Peripheral neuropathy; Taxanes; oxaliplatin; Chemotherapy; Venlafaxine
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Venlafaxine Hydrochloride; Gabapentin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Venlafaxine Arm (Experimental): Patients receiving Taxanes (Docetaxel or Paclitaxel) or Oxaliplatin containing regimens.
  Interventions: Drug: Venlafaxine 75 MG
- Gabapentin Arm (Active Comparator): Patients receiving Taxanes (Docetaxel or Paclitaxel) or Oxaliplatin containing regimens.
  Interventions: Drug: Gabapentin 400 mg

INTERVENTIONS:
Drug: Venlafaxine 75 MG — Venlafaxine 75 mg extended release capsules for a 7-days duration
  Arms: Venlafaxine Arm
Drug: Gabapentin 400 mg — Gabapentin 400 mg capsules
  Arms: Gabapentin Arm

SUMMARY:
Peripheral and Motor neuropathy represent a main obstacle for a better quality of life for cancer patients, Venlafaxine is introduced in a new dosing regimen for treating of oxaliplatin and taxanes induced peripheral neuropathy in cancer patients.

DETAILED DESCRIPTION:
Neurologic complications of anticancer therapy may result from direct toxic effects on the nervous system or via indirectly induced metabolic derangements or cerebrovascular disorders. A wide range of neurologic complications can associate antineoplastic drug treatment. Among the widely used anticancer drugs are the platinum-based compounds cisplatin and oxaliplatin which are the most commonly associated with various forms of neurotoxicity. Moreover, taxanes (paclitaxel) are also associated with neurotoxicity. In a double-blind trial in which 48 patients who treated with oxaliplatin-induced acute neurotoxicity were randomly assigned to venlafaxine (37.5 mg extended release twice daily from day 2 to 11) or placebo, however the 2014 systematic review of neuroprotectants from ASCO concluded that the venlafaxine data were not strong enough to recommend its use in clinical practice, until additional supporting data become available. patients will be randomly assigned to treatment arms:

1. Arm A: to receive venlafaxine hydrochloride 75 mg (Effexor X.R) 75mg once daily from day 1 to day 7 to avoid need of dose tapering .
2. Arm B: to receive Gabapentin 100-400 mg once daily from day 1 to day 7.

ELIGIBILITY:
Inclusion Criteria:

* Patients >24 years of age, men or women to lower risk of suicidal tendency.
* Patients with histologically proven cancer
* Patients receiving oxaliplatin or taxanes-based regimen
* WHO performance status of 0-2
* serum AST or ALT no higher than two times the upper limit of normal
* serum creatinine level less than 2 mg/dL
* platelet count of at least 100,000/mm3
* absolute neutrophil count of at least to 1.0 G/L
* Female patients, those with a negative urine pregnancy test.

Exclusion Criteria:

* Patients with brain or leptomeningeal metastasis.
* Patients with previous platinum-based chemotherapy
* Patients with history of alcoholic intoxication, diabetes, preexisting neuropathy or unstable psychological conditions.
* Patients with history of calcium/magnesium concomitant infusions, use of antiepileptics, antidepressants or lithium.

Ages: 24 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade II or more peripheral neuropathy | 4 months
  Grading of chemotherapy induced peripheral neuropathy will be done using NCI-CTCAE version (5)

SECONDARY OUTCOMES:
The EORTC QLQ-CIPN20 subscales | 4 months
  Sensory subscale, motor, and autonomic subscales of CIPN20
Pain Severity | 4 months
  The severity of neuropathic pain will be assessed using the Arabic version of the Brief Pain Inventory Short Form (BPI-SF)

CONTACTS AND LOCATIONS:
Locations (1):
- Mit Ghamr Oncology Center, Al Mansurah, Dakahlia Governorate, Egypt